CLINICAL TRIAL: NCT05771675
Title: Simvastatin Treatment to Improve Patient-reported Outcomes in Patients With Chronic Pancreatitis
Acronym: SMV in CP
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stephen Pandol, MD, Director, Basic and Translational Pancreas Research Medicine, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00002293
Record Dates: First submitted 2023-02-02; First posted 2023-03-16 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-04

CONDITIONS: Recurrent Acute Pancreatitis; Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis; Pancreatitis, Chronic | interventions — Simvastatin

STUDY DESIGN:
Intervention Model Description: Drug: Simvastatin Drug: Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Simvastatin (Experimental): Participants receive Simvastatin 40mg capsule once daily for 6 months.
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator): Participants receive Placebo capsule matching Simvastatin once daily for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — 40Mg Oral Tablet
  Arms: Simvastatin
Drug: Placebo — Matching Simvastatin Placebo tablet
  Arms: Placebo

SUMMARY:
The purpose of this pilot study to examine the feasibility and acceptability of simvastatin in adults with Recurrent Acute Pancreatitis (RAP) and Chronic Pancreatitis (CP).

DETAILED DESCRIPTION:
There are no available treatments for chronic pancreatitis (CP) or recurrent acute pancreatitis (RAP) and patients suffer with unremitting abdominal pain as the disease progress. This pilot study will test the feasibility of conducting a clinical trial of simvastatin to enhance the quality of life and delay disease progression in chronic pancreatitis patients. Emerging understanding of pancreas acinar cell organellar disorders underlying pancreatitis and the potential benefits of simvastatin to restore acinar cell homeostasis along with understanding of the pathways of the fibro-inflammatory response emanating from the disorders in the acinar cell allow the study team to propose a pilot placebo controlled double blind trial in patients with CP and RAP to test the effect of simvastatin on patient reported outcomes. Of note, RAP is a form of pancreatitis preceding CP.

The Study Team hypothesizes that treatment with simvastatin will have a significant benefit for reducing pain, improving health-related quality of life (HRQoL) and pancreatitis-related outcomes in patients with CP and RAP. Changes in blood biomarkers during treatments will provide biochemical evidence for the effectiveness of the treatments. The proposed study is a pilot double blind trial with 2:1 assignment of simvastatin vs placebo. 90 patients with either CP or RAP will be enrolled over a 24-month recruitment period. Treatment with simvastatin or placebo will be for 6 months. Outcome measures will be obtained at baseline, 3 months, and 6 months and 6 months after discontinuation of treatment for a total of one year. Feasibility and adherence will be monitored.

The Primary aim of this pilot study is to examine feasibility and acceptability of the trial in adults with RAP and CP. A priori thresholds to evaluate feasibility are: 50% enrollment, <15% attrition, >75% adherence with doses, <20% side effects, and >75% acceptability ratings. Multiple secondary outcome measures will be obtained that determine the effect of the treatments on pain and Quality of Life (QoL). The study plans to include male and female participants >18 years of age with Chronic and Recurrent Acute pancreatitis. Each participant will be involved for a period of 12 months from enrollment to completion of the study unless withdrawn by the study team for reasons of safety or by the participant for personal reasons.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18-75 at time of enrollment
4. Diagnosis of Recurrent Acute or Chronic Pancreatitis not attributable to gallstones (i.e., suspected or definite biliary etiology), medications, trauma or autoimmune pancreatitis. For CP, imaging studies that can be used for diagnosis classification using Cambridge criteria46,47.
5. Ability to take oral medication and be willing to adhere to the dosing regimen.
6. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional one month after administration of study medication.
7. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional one month after administration of study medication.
8. No prior pancreatic surgery
9. No current statin use for 6 months.

Exclusion Criteria:

1. Pregnancy or lactation
2. History of autoimmune, medication caused or traumatic pancreatitis.
3. Primary pancreatic tumors - pancreatic ductal adenocarcinoma, suspected cystic neoplasm (>1 cm. in size or main duct involvement), neuroendocrine tumors, and other uncommon tumors.
4. Pancreatic metastasis from other malignancies.
5. History of solid organ transplant, HIV/AIDS.
6. Known isolated pancreatic exocrine insufficiency (i.e.., in the absence of any eligible inclusion criteria).
7. Subjects required to take itraconazole, ketoconazole, erythromycin, clarithromycin, telithromycin, HIV protease inhibitors, nefazodone, gemfibrozil, cyclosporine, danazol, amiodarone, or verapamil for other clinical indications.
8. Current simvastatin use within the past 6 months.
9. Participants must not have medical or psychiatric illnesses or ongoing substance abuse that in the investigator's opinion would compromise their ability to tolerate study interventions or participate in longitudinal follow up.
10. Patients with active liver disease.
11. Known Pregnancy. All participants of childbearing potential, except if post-menopausal (i.e., no menses for ≥2 years) or had a hysterectomy, bilateral tubal ligation/clip (surgical sterilization) or surgical removal of both the ovaries), must have a negative urine or serum B-HCG pregnancy test documented within 2 days prior to any endoscopic or radiologic procedures done for research purposes. Any standard of care tests will follow institutional policies regarding pregnancy test.
12. Currently incarcerated.
13. Inability to comply with study activities.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Examine the feasibility and acceptability of testing the effect of simvastatin on health-related quality of life outcomes in patients with recurrent acute and chronic pancreatitis. | End of study (12 Months)
  A priori thresholds to evaluate feasibility are: 50% enrollment, <15% attrition, >75% adherence with doses, <20% side effects. A score of >75% acceptability ratings per an "Acceptability Form" that will be provided during the last visit will be used to gauge the general acceptability of the intervention (Simvastatin or Placebo) and study procedures to each participating subject.

SECONDARY OUTCOMES:
Determine the effect of simvastatin treatment on health-related quality of life (QoL) outcomes in patients with recurrent acute and chronic pancreatitis. | End of study (12 Months)
  Health-related quality of life measurements will be collected via questionnaires (PROMIS Sleep Disturbance and Physical Short Form, Physical Distress scale, pain scales, and the Pancreatic Quality of Life Instrument) to assess overall health, quality of life, and compare the mean change from baseline across the times points 3, 6, and 12 months between the treatment group and placebo in order to identify improvement in overall quality of life and pain management.
  The study will also collect blood samples to look for exploratory biomarkers to identify potential measures of response to treatment with the intent do develop larger efficacy focused trials.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Pandol, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: No